CLINICAL TRIAL: NCT01251692
Title: Ten-year Results of Phototherapeutic Keratectomy on Recurrent Corneal Erosions
Brief Title: Phototherapeutic Keratectomy (PTK) on Recurrent Corneal Erosions
Acronym: PTK x CE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Belquiz Rodrigues do Amaral Nassaralla, Instituto de Olhos de Goiânia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BQ-1-10-ARVO
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Recurrent Corneal Erosions
Keywords: Corneal erosions; PTK
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): A retrospective chart review of 26 eyes of 23 patients with recurrent corneal erosions treated by PTK from 1996 to 2000 was performed. All eyes had failed to respond to conventional therapy. Data regarding the preoperative and postoperative best-corrected visual acuity (BCVA), spherical equivalent (SE), symptomatic relief, incidence of recurrence, and complications arising from the laser treatment were analyzed. The mean duration of symptoms prior to PTK was 18 months (range, 8 to 36 months). The corneal epithelium was debrided, and laser ablation was performed to a depth of 5 micron with an ablation zone of 7 to 9 mm, using the Technolas 217C Plano Scan excimer laser. Mean postoperative follow-up was 12 years (range, 10 to 14 years).
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — The corneal epithelium was debrided, and laser ablation was performed to a depth of 5 micron with an ablation zone of 7 to 9 mm, using the Technolas 217C Plano Scan excimer laser.

SUMMARY:
To determine the ten-year visual results and outcome of excimer laser phototherapeutic keratectomy (PTK) for recurrent corneal erosions.

DETAILED DESCRIPTION:
A retrospective chart review of 26 eyes of 23 patients with recurrent corneal erosions treated by PTK from 1996 to 2000 was performed. All eyes had failed to respond to conventional therapy. Data regarding the preoperative and postoperative best-corrected visual acuity (BCVA), spherical equivalent (SE), symptomatic relief, incidence of recurrence, and complications arising from the laser treatment were analyzed. The mean duration of symptoms prior to PTK was 18 months (range, 8 to 36 months). The corneal epithelium was debrided, and laser ablation was performed to a depth of 5 micron with an ablation zone of 7 to 9 mm, using the Technolas 217C Plano Scan excimer laser. Mean postoperative follow-up was 12 years (range, 10 to 14 years).

ELIGIBILITY:
Inclusion Criteria:

Recurrent corneal erosions Patients 21 to 50 years old Conventional treatments have failed

Exclusion Criteria:

* Diabetes
* Autoimmune diseases

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 1996-01; Primary Completion 2000-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belquiz A Nassaralla, Study Chair — Instituto de Olhos de Goiânia